CLINICAL TRIAL: NCT04947501
Title: N9: Pilot Study of Novel Shortened Induction Chemotherapy for High-Risk Neuroblastoma
Brief Title: A Study of N9 Chemotherapy in Children With Neuroblastoma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-228
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Neuroblastoma; Pediatric Cancer
Keywords: HR-NB; Neuroblastoma; pediatric cancer; 21-228; Memorial Sloan Cancer Center
MeSH Terms: conditions — Neuroblastoma; Neoplasms | interventions — Cyclophosphamide; Topotecan; Vincristine; Doxorubicin; Ifosfamide; Etoposide; etoposide phosphate; Carboplatin; Mesna

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with newly-diagnosed HR-Neuroblastoma (Experimental): This pilot study of N9 as induction chemotherapy will enroll 30 patients with newly-diagnosed HR-NB. A first cohort of >1 to 12-year old, and a second cohort of extended age <19 years old. Both cohorts will be analyzed together.
  Interventions: Drug: Cyclophosphamide; Drug: Topotecan; Drug: Vincristine; Drug: Doxorubicin; Drug: Ifosfamide; Drug: Etoposide; Drug: Carboplatin; Drug: Mesna

INTERVENTIONS:
Drug: Cyclophosphamide — Administration of CTV - cycles 1 and 4
  Days 1 & 2: Cyclophosphamide 70 mg/kg/day (2100 mg/m2/day for patients >10 years old), IV over 6 hrs.
  Mesna 70 mg/kg (2100 mg/m2/day for patients >10 years old) , by 24-hr IV infusion, starting with the cyclophosphamide infusion.
  Days 1-4: Topotecan 2 mg/m2/day, IV over 30 minutes. Day 1: Vincristine 0.067 mg/kg (or 2 mg/m2, whichever is less) by IV piggyback; maximum dose is 2 mg.
  ******* Administration of CDV - cycle 3 Days 1 & 2: Cyclophosphamide 70 mg/kg/day ((2100 mg/m2/day for patients >10 years old), IV over 6 hrs.
  Mesna 70 mg/kg ((2100 mg/m2/day for patients >10 years old), by 24-hr IV infusion, starting with the cyclophosphamide infusion.
  Days 1-3: Doxorubicin 25 mg/m2/day, by 24-hr IV infusion (total dose over 72 hr is 75 mg/m2).
  Days 1-3: Vincristine 0.67 mg/m2/day or 0.022 mg/kg/day (whichever is less), by 24-hr IV infusion (total dose over 72 hr is 2 mg/m2 or 0.067 mg/kg); maximum dose is 0.67 mg/day, or 2mg over 72 hr.
  Other Names: Cytoxan
Drug: Topotecan — Administration of CTV - cycles 1 and 4
  Days 1 & 2: Cyclophosphamide 70 mg/kg/day (2100 mg/m2/day for patients >10 years old), IV over 6 hrs.
  Mesna 70 mg/kg (2100 mg/m2/day for patients >10 years old) , by 24-hr IV infusion, starting with the cyclophosphamide infusion.
  Days 1-4: Topotecan 2 mg/m2/day, IV over 30 minutes. Day 1: Vincristine 0.067 mg/kg (or 2 mg/m2, whichever is less) by IV piggyback; maximum dose is 2 mg.
  Other Names: Hycamtin
Drug: Vincristine — Administration of CTV - cycles 1 and 4
  Days 1 & 2: Cyclophosphamide 70 mg/kg/day (2100 mg/m2/day for patients >10 years old), IV over 6 hrs.
  Mesna 70 mg/kg (2100 mg/m2/day for patients >10 years old) , by 24-hr IV infusion, starting with the cyclophosphamide infusion.
  Days 1-4: Topotecan 2 mg/m2/day, IV over 30 minutes. Day 1: Vincristine 0.067 mg/kg (or 2 mg/m2, whichever is less) by IV piggyback; maximum dose is 2 mg.
  Other Names: Oncovin
Drug: Doxorubicin — Administration of CDV - cycle 3 Days 1 & 2: Cyclophosphamide 70 mg/kg/day ((2100 mg/m2/day for patients >10 years old), IV over 6 hrs.
  Mesna 70 mg/kg ((2100 mg/m2/day for patients >10 years old), by 24-hr IV infusion, starting with the cyclophosphamide infusion.
  Days 1-3: Doxorubicin 25 mg/m2/day, by 24-hr IV infusion (total dose over 72 hr is 75 mg/m2).
  Days 1-3: Vincristine 0.67 mg/m2/day or 0.022 mg/kg/day (whichever is less), by 24-hr IV infusion (total dose over 72 hr is 2 mg/m2 or 0.067 mg/kg); maximum dose is 0.67 mg/day, or 2mg over 72 hr.
  Other Names: Adriamycin
Drug: Ifosfamide — Administration of ICE - cycle 2 Days 1-5: Ifosfamide 1500 mg/m2/day (50 mg/kg/day if weight is <10 kg), IV over 6 hrs. Mesna 1500 mg/m2/day, by 24-hr IV infusion, starting with the ifosfamide infusion. Days 1-2: Carboplatin 400 mg/m2/day (13.3 mg/kg/day if weight is <10 kg), IV over 1 hr. Days 1-5: Etoposide 100 mg/m2/day (3.3. mg/kg/day if weight is <10 kg), IV over 2 hrs.
  Other Names: Isophosphamide
Drug: Etoposide — Administration of ICE - cycle 2
  Days 1-5: Ifosfamide 1500 mg/m2/day (50 mg/kg/day if weight is <10 kg), IV over 6 hrs. Mesna 1500 mg/m2/day, by 24-hr IV infusion, starting with the ifosfamide infusion. Days 1-2: Carboplatin 400 mg/m2/day (13.3 mg/kg/day if weight is <10 kg), IV over 1 hr. Days 1-5: Etoposide 100 mg/m2/day (3.3. mg/kg/day if weight is <10 kg), IV over 2 hrs.
  Other Names: VePesid; Etopophos
Drug: Carboplatin — Administration of ICE - cycle 2
  Days 1-5: Ifosfamide 1500 mg/m2/day (50 mg/kg/day if weight is <10 kg), IV over 6 hrs. Mesna 1500 mg/m2/day, by 24-hr IV infusion, starting with the ifosfamide infusion. Days 1-2: Carboplatin 400 mg/m2/day (13.3 mg/kg/day if weight is <10 kg), IV over 1 hr. Days 1-5: Etoposide 100 mg/m2/day (3.3. mg/kg/day if weight is <10 kg), IV over 2 hrs.
  Other Names: Paraplatin
Drug: Mesna — Administration of CTV - cycles 1 and 4 Mesna 70 mg/kg (2100 mg/m2/day for patients >10 years old) , by 24-hr IV infusion, starting with the cyclophosphamide infusion.
  Administration of ICE - cycle 2 Mesna 1500 mg/m2/day, by 24-hr IV infusion, starting with the ifosfamide infusion.
  Administration of CDV - cycle 3 Mesna 70 mg/kg ((2100 mg/m2/day for patients >10 years old), by 24-hr IV infusion, starting with the cyclophosphamide infusion.
  Other Names: Mesnex

SUMMARY:
The purpose of the study is to find out whether N9 is a safe and effective treatment for children with neuroblastoma. N9 includes 3 different combinations of chemotherapy drugs that are given at different times - Cyclophosphamide, topotecan, and vincristine (CTV), Ifosfamide, carboplatin, and etoposide (ICE), Cyclophosphamide, doxorubicin, and vincristine (CDV).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NB as defined by histopathology (confirmed by the MSK Department of Pathology), BM metastases plus high urine catecholamine levels, or positivity in MIBG scan.
* HR-NB, defined as MYCN-amplified stage 2/3/4/4S at any age and stage 4 in patients >18 months old.
* No more than one prior cycle of chemotherapy.
* Age <19 years old.
* Signed informed consent indicating awareness of the investigational nature of this treatment.

Exclusion Criteria:

* Severe dysfunction of major organs, i.e., renal, cardiac, hepatic, neurologic, pulmonary, hematologic, or gastrointestinal toxicity ≥ grade 3.
* Inability to comply with protocol requirements.
* Pregnancy is not an issue because all patients will be pre-adolescents.

Ages: 1 Year to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2026-06-22 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Assess safety of the N9 regimen in participants with HR-NB through toxicity assessment | 16 weeks
  Adverse events will be graded using Common Toxicity Criteria Version 5.0 developed by the National Cancer Institute of the USA, events of all grades will be tabulated, for non-hematologic effects and hematologic effects on the patients in the safety set. The timing of cycles will also be described to assess any delay due to toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kushner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org